## **DATA ANALYSIS 29/9/17**

## Patient morbidity after palatal free gingival grafts with or without PRF membranes coverage: a comparative randomized clinical trial.

F. Gatti<sup>1</sup>, E. Scaramuzza<sup>1</sup>, M.Chiapasco<sup>2</sup>

<sup>&</sup>lt;sup>1</sup> Unit of Oral Surgery (Head Prof. Matteo Chiapasco) - Department of Health Sciences – San Paolo Hospital, University of Milan, Italy

<sup>&</sup>lt;sup>2</sup>Head Unit of Oral Surgery - Department of Health Sciences – San Paolo Hospital, University of Milan, Italy

## Data analysis

A statistical application (SPSSS Windows 18.0, Chicago; IL, USA) was used for the statistical analysis by a blind operator.

The patient was the statistical unit of this analysis.

T-test for indipendent samples was used to evaluate differences between the test and the control group regarding the mean consumption of pain killers (mg).

Mann-Whitney U test was used to compare medians of the two groups for the following parameters: post-surgical pain related to donor site and grafting site (VAS), post-operative discomfort (VAS), inability to chew (VAS), stress (VAS) and post-surgical bleeding (VAS).

Furthermore, median and values of interquartiles (IRQ) were calculated for a better description of the presented datas.

A statistically significant difference was defined as p < 0.05.